CLINICAL TRIAL: NCT02723968
Title: Sensitivity and Specificity of Different Methods for Cystic Fibrosis-related Diabetes Screening.
Brief Title: Cystic Fibrosis Related Diabetes Screening.
Acronym: D2M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008.527
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-03

CONDITIONS: Cystic Fibrosis-related Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous glucose monitoring system (Other): OGTT followed by continuous glucose monitoring system and finally IGTT and HbA1C dosage
  Interventions: Other: glucose solution at a dose of 1.75 g/kg (up to a maximum of 75 g) for the OGTT and glucose solution at a dose of 0.5 g/kg (up to a maximum of 35 g) was injected in 2.5-3 min for the IGTT; Procedure: HGPIV diagnosis test; Procedure: HOMAR-IR diagnosis test

INTERVENTIONS:
Other: glucose solution at a dose of 1.75 g/kg (up to a maximum of 75 g) for the OGTT and glucose solution at a dose of 0.5 g/kg (up to a maximum of 35 g) was injected in 2.5-3 min for the IGTT — At the first visit at day 1an OGTT will be performed then the CGMS is implanted. Capillary glycaemia will be taken four times a day to set up the CGMS. A second visit is scheduled at day 4, where the intravenous glucose tolerance test is performed as well as the HbA1C level.
Procedure: HGPIV diagnosis test
Procedure: HOMAR-IR diagnosis test

SUMMARY:
Cystic fibrosis-related diabetes is a late cystic fibrosis (CF) associated comorbidity whose prevalence is increasing sharply lifelong. Guidelines for glucose metabolism (GM) monitoring relies on oral glucose tolerance test . However, this test is neither sensitive nor specific.

The aim of this study is to compare sensitivity and specificity of different methods for GM monitoring in children and adolescents with CF.

Continuous GM system (CGMS) will be used as the reference method. Results will be compared to those of oral glucose tolerance test (OGTT), intravenous glucose tolerance test (IGTT), homeostasis model assessment index of insulin resistance (HOMA-%IR) , homeostasis model assessment index of beta-cell function (HOMA-%B) and HbA1C dosage (glycated haemoglobin A1C). Patients will be classified into three groups according to CGMS: normal glucose tolerance, impaired glucose tolerance and diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of Cystic Fibrosis with a sweat chloride > 60 mmol/L.
* Subjects will be aged between 10 and 18 years with at least one class 1 or 2 Cystic fibrosis transmembrane conductance regulator (CFTR) mutation.
* Subjects will be pancreatic insufficient.
* Subjects must have a forced expiratory volume 1 (FEV1)> 40 % of predicted normal for age, sex and height at the screening visit.
* Stable CF disease as judged by the investigator

Exclusion Criteria:

* Subjects with glucose intolerance abnormalities
* Subjects with pulmonary exacerbation within 4 weeks before screening
* History of lung or hepatic transplantation or awaiting transplantation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the sensitivity and the specificity of IGTT (intravenous glucose tolerance test) for the diagnosis of diabetes mellitus in comparison to a continuous glucose monitoring system | Day 3
Measurement of the sensitivity and the specificity of HOMA-%IR (homeostasis model assessment index of insulin resistance) for the diagnosis of diabetes mellitus in comparison to a continuous glucose monitoring system. | Day 3

SECONDARY OUTCOMES:
Measurement of the prevalence of diabetes mellitus. | Day 3
Correlation between IGTT and HOMA-%IR data and HbA1C dosage (glycated haemoglobin A1C). | Day 3
Measurement of glucose intolerance | Day 3
Correlation between IGTT and HbA1C dosage (glycated haemoglobin A1C). | Day 3

REFERENCES:
- [Result] Mainguy C, Bellon G, Delaup V, Ginoux T, Kassai-Koupai B, Mazur S, Rabilloud M, Remontet L, Reix P. Sensitivity and specificity of different methods for cystic fibrosis-related diabetes screening: is the oral glucose tolerance test still the standard? J Pediatr Endocrinol Metab. 2017 Jan 1;30(1):27-35. doi: 10.1515/jpem-2016-0184. PMID 27977404